CLINICAL TRIAL: NCT05542563
Title: The Influence of Mindfulness on Patient-Reported Outcomes, Return to Sport and Re-Injury Following Anterior Cruciate Ligament (ACL) Reconstruction Surgery
Brief Title: Mindfulness and ACL Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0845; Protocol Version 10/10/2023 (Other: UW Madison); A536110 (Other: UW Madison)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: ACL; ACL Injury
Keywords: ACL Surgery; mindfulness
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: a single-blind, randomized controlled trial design to evaluate the effects of a remotely-delivered 8-week mindfulness intervention on patient-reported outcomes following ACL reconstruction surgery
Who Masked: Care Provider
Masking Description: All healthcare providers involved in the care of the participant following surgery (surgeon, physician's assistants, nurses, medical assistants, etc.) will be blinded to the group assignment of each participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention plus Standard of Care (Experimental): The Foundations and Awareness modules of the HMP app require a minimum of 133 and 253 minutes, equating to less than 5 and less than 10 minutes per day on average, respectively. Date, duration, and content of usage will be recorded for each participant through the app. Participants will have access to the entire contents of the app for the full duration of the study.
  Interventions: Behavioral: Healthy Minds Program (HMP) App
- Standard of Care (No Intervention): Control group receives standard of care only

INTERVENTIONS:
Behavioral: Healthy Minds Program (HMP) App — The full HMP app includes 5 modules with practices designed to cultivate categories of mental and emotional skills linked to both hedonic and eudaimonic well-being. These include the cultivation of mindful attention (Awareness), positive relationships with self and others (Connection), insight into the nature of self and internal experience (Insight), and purpose, values, and meaning in life (Purpose), as well as an initial module which includes abbreviated introductions to the topics and lessons in all four areas (Foundations). For this study, the active intervention will include 4 weeks of training using the Foundations module followed by 4 weeks of training using the Awareness module.
  Arms: Mindfulness Intervention plus Standard of Care

SUMMARY:
Anterior cruciate ligament (ACL) surgery patients experience physical trauma, both in the physical injury itself and following surgery, and face potential long-lasting adverse effects such as muscle weakness, diminished joint function, hip pain, and fear. Many of these patients report more significant anxiety and depression following surgery, which can further compound these patients' adverse outcomes. This study is a single-blind, randomized controlled trial design to evaluate the effects of a remotely-delivered 8-week mindfulness intervention on patient-reported outcomes (PROs) following ACL reconstruction surgery.

DETAILED DESCRIPTION:
Rationale and Approach: ACL reconstruction surgery patients experience physical trauma, both in the physical injury itself and following surgery, and face potential adverse long-lasting effects such as muscle weakness, arthritis, persistent knee pain, anxiety, depression, post-traumatic stress, and fear of re-injury. Many of these patients report sufficient psychological trauma that undermines a return to sport and potentially contributes to the risk of re-injury to the repaired knee. This study is a single-blind, randomized controlled trial design to evaluate the effects of a remotely-delivered 8-week mindfulness intervention on patient-reported outcomes following ACL reconstruction surgery.

* Specific Aim 1: To determine the influence of mindfulness training on patient-reported outcomes and return to sport following ACL reconstruction surgery

  * Hypothesis 1: Mindfulness training will be associated with improvements in pain, quality of life, depression, anxiety, post-traumatic stress and fear of re-injury, as well as greater likelihood of returning to sport in the 24 months following ACL reconstruction surgery
* Specific Aim 2: To determine the influence of mindfulness training on re-injury risk following ACL reconstruction surgery

  * Hypothesis 2: Among those participants that return to sport, mindfulness training will be associated with a decreased risk of ipsilateral ACL rupture in the 24 months following ACL reconstruction surgery
* Specific Aim 3: To determine the factors that influence mindfulness efficacy in patient-reported outcomes and return to sport following ACL reconstruction surgery

  * Hypothesis 3: Among participants in the mindfulness group, total duration of mindfulness training and female gender will be independently associated with improvements in pain, quality of life, depression, anxiety, post-traumatic stress and fear of re-injury, as well as greater likelihood of returning to sport in the 24 months following ACL reconstruction surgery

ELIGIBILITY:
Inclusion Criteria:

* 16-40 years old at the time of the pre-operative visit
* Regular access to a mobile device compatible with the Healthy Minds Program (HMP) App (Android or iOS)
* Undergoing ACL surgery

Exclusion Criteria:

* Prior diagnosis of serious mental illness (schizophrenia, bipolar disorder, schizoaffective disorder, etc).
* Significant prior experience with meditation or mindfulness, defined as greater than 30 minutes in a month during the past year
* Knee injury requiring multi-ligament reconstruction
* Prior ipsilateral knee surgery
* Prior contralateral ACL reconstruction

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS Global Health Questionnaire (GHQ) Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Global quality of life (QoL) will be assessed via a 9-item questionnaire scored on a 0-100 scale where higher scores indicate better QoL, pain interference, and fatigue.
Change in PROMIS Anxiety Questionnaire Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Anxiety will be assessed via an 8-item questionnaire scored from 0-5 where higher scores represents greater anxiety.
Change in PROMIS Depression Questionnaire Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Depression will be assessed via an 8-item questionnaire scored from 0-5 where higher scores represents greater depression.
Change in Single Assessment Numeric Evaluation (SANE) Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Pain severity is assessed via a single item survey scored from 0-100 where a higher score indicates greater pain.
Change in Horowitz Impact of Events Scale Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Post-traumatic stress is assessed via a 15-item survey scored from 0-3 where higher scores indicate greater level of post-traumatic stress.
Change in Tampa Scale of Kinesiophobia 11 (TSK-11) Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Fear of re-injury is assessed via an 11-item survey scored from 1-4 where higher scores indicate a greater fear of re-injury.
Change in Pain Catastrophizing Scale (PCS) Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Pain catastrophizing is assessed via a 13-item survey scored from 0-4 where higher scores indicate a higher level of pain catastrophizing.
Change in Anterior Cruciate Ligament Return to Sport After Injury scale (ACL-RSI) Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Psychological readiness is assessed via a 12-item survey scored on an 11-point scale where higher scores indicate a higher level of readiness.
Change in Athletic Identity Measurement Scale (AIMS) Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Athletic identity is assessed via a 10-item survey with a total range of scores from 10-70 where higher scores indicate a higher level of athletic identity.
Change in International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form Score | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Knee function is assessed via a 10-item survey scored from 0-10 where higher scores means less limitation with activities and less symptoms.
Change in General physical activity questionnaire (GPAQ) Measured as Minutes of Total Physical Activity per day | baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Higher score indicates higher physical activity.

SECONDARY OUTCOMES:
Knee Range of Motion | 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
Peak Torque | 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Participants will undergo testing of resisted flexion and extension to determine peak torque
Peak Torque Relative to Body Weight | 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Participants will undergo testing of resisted flexion and extension to determine peak torque relative to body weight
Hamstring to Quadriceps Torque Ratio | 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  Participants will undergo testing of resisted flexion and extension to determine hamstring to quadriceps torque ratio.
Change in Jump Landing Assessment: Force Measures | 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  loading force, acceleration force, landing force, peak landing force on both legs together
Change in Jump Height | 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
Change in Vertical Hop Testing: Force Measures | 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
  down force, up force, landing force, peak landing force on a single leg
Change in Hop Height | 6 weeks, 3 months, 6 months, 12 months, 24 months post surgery
Total Duration of Mindfulness Intervention in the Mindfulness Group | up to 24 months
Number of Participants Who Return to Sport | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Watson, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No